CLINICAL TRIAL: NCT05336721
Title: An Open Labelled, Multicenter-phase II Study of Chiauranib Combine With Capecitabine in Advanced Triple-negative Breast Cancer Failed to Prior Anthracyclines and Taxanes Therapy
Brief Title: A Phase II Study of Chiauranib in Combine With Capecitabine in TNBC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: During the enrollment period of this project, due to the increasing proportion of patients receiving capecitabine adjuvant therapy and the large number of trials competing for the same number of lines in various centers
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR202
Record Dates: First submitted 2022-04-14; First posted 2022-04-20 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-11

CONDITIONS: Triple-negative Breast Cancer
Keywords: Chiauranib；Capecitabine；triple-negative breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — chiauranib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Chiauranib + capecitabine (Experimental): Patients receive the combined treatment of Chiauranib plus capecitabine, 21 days as a cycle until objective disease progression.
  Interventions: Drug: Chiauranib; Drug: capecitabine

INTERVENTIONS:
Drug: Chiauranib — 25mg/35mg/50mg orally once daily
Drug: capecitabine — 1000mg/m2 on Days 1-14 in a repeating 21-day cycle

SUMMARY:
This study is to evaluate the preliminary efficacy and safety of chiauranib in combine with capecitabine in advanced triple-negative breast cancer failed to prior anthracyclines and taxanes therapy

DETAILED DESCRIPTION:
Chiauranib is a novel orally active multi-target inhibitor that simultaneously inhibits the angiogenesis-related kinases (VEGFR2, VEGFR1, VEGFR3,PDGFRa and c-Kit), mitosis-related kinase Aurora B and chronic inflammationrelated kinase CSF-1R in a high potency manner with the IC50 at a single-digit nanomolar range. In particular, Chiauranib showed very high selectivity in the kinase inhibition profile with little activity on off-target nonreceptor kinases, proteins, GPCR and ion channels, indicative of a better drug safety profile in terms of clinical relevance.

This study including two phases: (1) dose-escalation , this phase using a 3+3design，9-18 patients will be enrolled and receive 25mg/35mg/50mg chiauranib and 1000mg/m2 capecitabine Q3W. (2) dose-expansion，About 20 patients will be enrolled and receive the MTD dose of chiauranib and 1000mg/m2 capecitabine Q3W.

This study also to explore the PK variation and gene expression via blood samples

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have given signed, informed consent prior to registration on study
2. age ≥ 18 years
3. female
4. Histological or cytological evidence of estrogen-receptor negative (ER-), progesterone receptor negative (PgR-) and human epidermal growth factor-2 receptor negative (HER2-) Breast Cancer by local laboratory testing.
5. Patients with locally advanced inoperable or recurrent/metastatic TNBC and had failed treatment with anthracyclines and taxanes.
6. At least 1 lesion can be accurately measured, as defined by RECIST1.1
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
8. Laboratory criteria are as follows:

1) Complete blood count: hemoglobin (Hb) ≥90g/L ; absolute neutrophil count (ANC) ≥1.5×109/L ; platelets ≥90×109/L; 2) Biochemistry test: serum creatinine(cr) <1.5×ULN; total bilirubin<1.5×ULN; alanine aminotransferase(ALT) ,aspartateaminotransferase(AST)≤2.5×ULN; (ALT,AST#5×ULN if liver involved) 3) Coagulation test: International Normalized Ratio (INR) < 1.5

9. Life expectancy of at least 3 months

Exclusion Criteria:

1. Patients have used any anti-cancer therapy, including adiotherapy, chemotherapy, immunotherapy, target therapy, and other anti-tumor treatments within 28 days before the first dose
2. Patients received vascular endothelial growth factor(VEGF)/vascular endothelial growth factor receptor(VEGFR) inhibitor, like Apatinib, Anlotinib, Fruquintinib, Bevacizumab, etc., or Aurora kinase inhibitors, etc; Patients had treatment of capecitabine (except who received the treatment of capecitabine in Neoadjuvant/ Adjuvant therapy, and Recurrence occurs after 12 months)
3. Has known allegies to Chiauranib, capecitabine or any of the excipients
4. prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer
5. Treatment with an investigational agent/instrument within 28 days prior to first dose of study drug
6. Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1
7. Patients with prior invasive malignancies in the past five years with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or cervical carcinoma in situ
8. History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis
9. Have uncontrolled or significant cardiovascular disease, including:

1) Congestive heart failure, unstable angina pectoris, myocardial infarction within 6 months prior to study entry; arrhythmia, or Left Ventricular Ejection Fraction (LVEF) < 50% requiring treatment with agents during screening stage 2) primary cardiomyopathy(dilated cardiomyopathy, hypertrophic cardiomyocyte, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, et,al) 3) History of significant QT interval prolongation, or Corrected QT Interval (QTc) > 470 ms prior to study entry 4) Symptomatic coronary heart disease requiring treatment with agents 5) History of hypertension treated by≥2 agents, or the Blood pressure(Bp) ≥140/90 mmHg prior to study entry 6) Other condition investigator considered inappropriate

10. CT or MRI of the chest during the screening period shows interstitial lung disease or pulmonary fibrosis or lung inflammation that requires treatment, or within 6 months before the first dose, history of pneumonia requiring oral or intravenous steroid treatment

11. Have clinical significant gastrointestinal abnormality that would impair the ingestion, transportation or absorption of oral agents, history of gastrointestinal perforation or abdominal fistula, peptic ulcer disease within 6 months prior to first dose of study drug

12. Urinary protein ≥ 2+ and quantitative urinary protein ≥ 1g/24 h during the screening period

13. History of active bleeding within the past 2 months, patients with bleeding potential during the screening period, or receiving anticoagulation therapy

14. Pleural fluid, ascites or pericardial effusion with significant symptoms or required treatment of puncture or drainage during the screening period

15. History of deep venous thrombosis or Pulmonary embolism within the past 6 months

16. Active infection requiring oral or intravenous systemic antimicrobial therapy during the screening period

17. Screening for HIV antibody positive

18. Screening test for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive with virus replication, hepatitis C antibody (HCVAb) positive with virus replication

19. Any mental or cognitive disorder, that would impair the ability to understand the informed consent document, or the compliance of study

20. Candidates with drug and alcohol abuse

21. Participants of reproductive potential not willing to use adequate contraceptive measures for the duration of the study.Pregnant or breastfeeding women

22. Any other condition which is inappropriate for the study in the opinion of the investigators

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
ORR(Objective reponse rate) | 2years
  Overall response rate (ORR) is defined as the percentage of patients with complete or partial response evaluated by RECIST 1.1. Per RECIST 1.1: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR

SECONDARY OUTCOMES:
CBR (Clinical Benefit Rate) | 2years
  Clinical Benefit Rate (CBR) will be determined by looking at the number of subjects who have either a complete response, partial response, or stable disease for greater than or equal to 24 weeks, per RECIST 1.1
PFS (Progression-free survival) | 2years
  From date of the first dose of study drug until the date of first documented progression or relapse or date of death from any cause, whichever came first,
DoR (Duration of response) | 2years
OS(Overall survival) | 2years
AEs | 2years
  percentage of AEs

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No